CLINICAL TRIAL: NCT03092765
Title: A Clinical Phase 2 Study of E6011 in Japanese Subjects With Primary Biliary Cholangitis Inadequately Responding to Ursodeoxycholic Acid
Brief Title: Study of E6011 in Japanese Subjects With Primary Biliary Cholangitis Inadequately Responding to Ursodeoxycholic Acid
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision (non-safety related)
Sponsor: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E6011/ET1
Record Dates: First submitted 2017-03-24; First posted 2017-03-28 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-07

CONDITIONS: Primary Biliary Cholangitis
Keywords: E6011; Ursodeoxycholic acid; Japan
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — quetmolimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- low-dose, high-frequency E6011; high-dose, low-frequency E6011 (Experimental): Participants will receive low-dose E6011 at a relatively higher frequency up to approximately Week 12. Participants will then receive high-dose E6011 at a relatively lower frequency from Week 12 to Week 64.
  Interventions: Drug: E6011
- low-dose, high-frequency E6011; low-dose, low-frequency E6011 (Experimental): Participants will receive low-dose E6011 at a relatively higher frequency up to approximately Week 12. Participants will then receive low-dose E6011 at a relatively lower frequency from Week 12 to Week 64.
  Interventions: Drug: E6011
- high-dose, low-frequency E6011; high-dose, low-frequency E6011 (Experimental): Participants will receive high-dose E6011 at a relatively lower frequency up to approximately Week 12. Participants will then receive high-dose E6011 at a relatively lower frequency from Week 12 to Week 64.
  Interventions: Drug: E6011
- high-dose, low-frequency E6011; low-dose, low-frequency E6011 (Experimental): Participants will receive high-dose E6011 at a relatively lower frequency up to approximately Week 12. Participants will then receive low-dose E6011 at a relatively lower frequency from Week 12 to Week 64.
  Interventions: Drug: E6011
- low-dose, low-frequency E6011; high-dose, low-frequency E6011 (Experimental): Participants will receive low-dose E6011 at a relatively lower frequency up to approximately Week 12. Participants will then receive high-dose E6011 at a relatively lower frequency from Week 12 to Week 64.
  Interventions: Drug: E6011
- low-dose, low-frequency E6011; low-dose, low-frequency E6011 (Experimental): Participants will receive low-dose E6011 at a relatively lower frequency up to approximately Week 12. Participants will then receive low-dose E6011 at a relatively lower frequency from Week 12 to Week 64.
  Interventions: Drug: E6011
- Placebo; high-dose, low-frequency E6011 (Experimental): Participants will receive placebo up to approximately Week 12. Participants will then receive high-dose E6011 at a relatively lower frequency from Week 12 to Week 64.
  Interventions: Drug: E6011; Drug: Placebo
- Placebo; low-dose, low-frequency E6011 (Experimental): Participants will receive placebo up to approximately Week 12. Participants will then receive low-dose E6011 at a relatively lower frequency from Week 12 to Week 64.
  Interventions: Drug: E6011; Drug: Placebo

INTERVENTIONS:
Drug: E6011 — Intravenous administration
Drug: Placebo — Intravenous administration
  Arms: Placebo; high-dose, low-frequency E6011; Placebo; low-dose, low-frequency E6011

SUMMARY:
This study is a placebo-controlled, randomized, double-blind, multicenter, parallel-group comparison study in primary biliary cholangitis participants inadequately responding to ursodeoxycholic acid.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary biliary cholangitis corresponding to one of the following criteria:

  * Histologically confirmed chronic non-suppurative destructive cholangitis (CNSDC) with laboratory findings compatible with primary biliary cholangitis (PBC)
  * Positivity for antimitochondrial antibodies (AMAs) with histological findings compatible with PBC but in the absence of characteristic histological findings of CNSDC
  * No histological findings available, but positivity for AMAs as well as clinical findings and a course indicative of typical cholestatic PBC
* Aged ≥20 and <75 years old at the time of informed consent
* Taking stable dose of ursodeoxycholic acid for at least 6 months (≥600 milligrams [mg]/day) prior to Screening
* Screening and Week 0 alkaline phosphatase (ALP) values between 1.67 and 10 times the upper limit of normal
* Outpatient
* Has voluntarily consented, in writing, to participate in this study, and is able to comply with all aspects of the protocol

Exclusion Criteria:

* Received the following drugs within 12 weeks before starting the study treatment:

  * Drugs that suppose the efficacy to PBC:

    o azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate mofetil, penicillamine, fibrates, and other systemic corticosteroids
  * Potentially hepatotoxic drugs o methyl-dopa, sodium valproic acid, and isoniazide
* History or current condition of hepatic decompensation with variceal bleeds, encephalopathy ≥ grade 2 and poorly controlled ascites, and history of liver transplantation
* History or current condition of other concomitant liver diseases including hepatitis due to hepatitis B virus (HBV)/hepatitis C virus (HCV) infection, primary sclerosing cholangitis, alcoholic liver disease (including liver cirrhosis), autoimmune liver disease requiring the treatment of systemic corticosteroids or biopsy proven non-alcoholic steatohepatitis (NASH)
* History or current clinical condition of malignant tumor, lymphoma, leukemia, or lymphoproliferative disease, except for skin carcinoma (epithelial carcinoma or basal cell carcinoma) and cervix carcinoma which has completely excised and without metastasis or recurrence for more than 5 years before informed consent
* Immunodeficiency or history of human immunodeficiency virus (HIV) infection
* Infection requiring hospitalization or intravenous administration of antibiotics or disease requiring administration of antivirus drugs (eg, herpes zoster) within 4 weeks before starting the study treatment
* History of tuberculosis or current complication of active tuberculosis
* Positive tuberculosis test (QuantiFERON®TB Gold Test or T-SPOT®.TB Test) at Screening
* History of clinically important vasculitis
* History of severe allergy (shock or anaphylactoid symptoms)
* Complication of uncontrolled disorders such as acute cardiac infarction, unstable angina, brain infarct, or symptomatic intracerebral hemorrhage
* Evidence of clinically significant disease (eg, cardiac, respiratory, gastrointestinal, or renal disease) that could affect the participant's safety or interfere with the study assessments in the opinion of the investigator or subinvestigator
* Tested positive for any of the following at Screening: HIV, hepatitis B surface (HBs) antigen, HBs antibody, hepatitis B core (HBc) antibody, HBV deoxyribonucleic acid (DNA), HCV antibody, human T-lymphotropic virus type 1 (HTLV-1) antibody, or syphilis
* Demonstrated prolonged QT interval corrected using Fridericia's formula (QTcF) interval (>450 milliseconds [ms]) in repeated electrocardiogram examinations
* Received immunoglobulin preparations or blood products within 24 weeks before starting the study treatment
* Received a live vaccine within 12 weeks before starting the study treatment, or is planning to receive
* Females who are, or may be pregnant, who are breastfeeding, who wish to become pregnant during the study period, and females or their partners who do not wish to use reliable contraceptive measures.
* Scheduled for surgery before Week 64
* Has been treated with investigational drugs in other E6011 study
* Currently enrolled in another clinical study, including the follow-up
* Used any investigational drug within 28 days (or 5× the half-life, whichever is longer) before informed consent
* Judged to be ineligible to participate in this study by the investigator or sub-investigator

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Rate of change from Baseline in serum alkaline phosphatase (ALP) values at Week 12 | Baseline; Week 12
  This assessment will be conducted as a measure of efficacy.

SECONDARY OUTCOMES:
Number of participants with a decrease in ALP response rates of 15%, 20%, and 40% from Baseline | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Number of participants with an ALP value less than 1.67 times the upper limit normal and a total bilirubin value within normal limits and a greater than or equal to 15% decrease in ALP from Baseline | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean values of serum ALP, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean values of gamma-guanosine-5'-triphosphate (γGTP) at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean values of serum total bilirubin and direct bilirubin at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean values of serum total bile acids at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean values of serum albumin at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean change from Baseline in serum ALP, AST, and ALT at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean change from Baseline in serum γGTP at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean change from Baseline in serum total bilirubin and direct bilirubin at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean change from Baseline in serum total bile acids at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean change from Baseline in serum albumin at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean rate of change from Baseline in serum ALP, AST, and ALT at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean rate of change from Baseline in serum γGTP at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean rate of change from Baseline in serum total bilirubin and direct bilirubin at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean rate of change from Baseline in serum total bile acids at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean rate of change from Baseline in serum albumin at each visit | Baseline; up to Week 64
  This assessment will be conducted as a measure of efficacy.
Mean change from Baseline in individual domain and total primary biliary cholangitis (PBC) version Child-Pugh scores | Screening; up to Week 64
  The Child-Pugh classification is used to assess the prognosis of chronic liver disease. The score employs five clinical measures of liver disease. Each measure is scored from 1 to 3, with 3 indicating most severe derangement. The total score ranges from 5 to 15 and is a sum of the individual domain scores. A higher score indicates a worse prognosis.
Mean change from Baseline in domain (Symptoms, Itch, Fatigue, Cognitive, Emotional, Social) and total scores on the PBC-40 | Baseline; up to Week 64
  The PBC-40 is measures quality of life. Participants are asked to respond to 40 questions, each of which is scored on a scale of 0 to 5 (where 0=not applicable; 1=least impact; 5=greatest impact), grouped into six domains (symptoms, itch, fatigue, cognition, social, and emotional). For each domain, scoring involves summing individual question response scores. A higher score indicates a poorer quality of life.
Mean change from Baseline in each score (fibrosis, bile duct loss, deposition of orcein-positive granules) and total scores, in the stage based on the total scores, in each score of cholangitis activity and hepatitis activity on Nakanuma classification | Screening; Weeks 52 to 60
  Scores for fibrosis, bile duct loss, and chronic cholestasis are combined for staging: stage 1, total score of 0; stage 2, score 1 to 3; stage 3, score 4 to 6; and stage 4, score 7 to 9. Cholangitis activity and hepatitis activity are graded as CA0-3 and HA0-3, respectively. A higher score indicates more severe disease.
Mean values of fibrosis marker at each visit | Baseline; up to Week 64
  The presence of serum fibrosis markers may be correlated with PBC.
Mean change from Baseline in fibrosis marker at each visit | Baseline; up to Week 64
  The presence of serum fibrosis markers may be correlated with PBC.
Mean rate of change from Baseline in fibrosis marker at each visit | Baseline; up to Week 64
  The presence of serum fibrosis markers may be correlated with PBC.
Mean values of fibrosis 4 (Fib-4) index at each visit | Baseline; up to Week 64
  The presence of serum fibrosis markers may be correlated with PBC.
Mean change from Baseline in Fib-4 index at each visit | Baseline; up to Week 64
  The presence of serum fibrosis markers may be correlated with PBC.
Mean rate of change from Baseline in Fib-4 index at each visit | Baseline; up to Week 64
  The presence of serum fibrosis markers may be correlated with PBC.

CONTACTS AND LOCATIONS:
Locations (46):
- Japan (46):
  - EA Pharma trial site, Nagoya, Aichi-ken
  - EA Pharma trial site, Matsudo, Chiba
  - EA Pharma trial site, Touon, Ehime
  - EA Pharma trial site, Yoshida, Fukui
  - EA Pharma trial site, Kurume, Fukuoka
  - EA Pharma trial site, Maebashi, Gunma
  - EA Pharma trial site #1, Sapporo, Hokkaido
  - EA Pharma trial site #2, Sapporo, Hokkaido
  - EA Pharma trial site, Kobe, Hyōgo
  - EA Pharma trial site, Nishinomiya, Hyōgo
  - EA Pharma trial site, Inashiki, Ibaraki
  - EA Pharma trial site, Morioka, Iwate
  - EA Pharma trial site, Kita, Kagawa-ken
  - EA Pharma trial site, Takamatsu, Kagawa-ken
  - EA Pharma trial site #1, Yokohama, Kanagawa
  - EA Pharma trial site #2, Yokohama, Kanagawa
  - EA Pharma trial site, Sendai, Miyagi
  - EA Pharma trial site, Matsumoto, Nagano
  - EA Pharma trial site, Oomura, Nagasaki
  - EA Pharma trial site, Kashihara, Nara
  - EA Pharma trial site, Nakagami, Okinawa
  - EA Pharma trial site, Hirakata, Osaka
  - EA Pharma trial site #1, Suita, Osaka
  - EA Pharma trial site #2, Suita, Osaka
  - EA Pharma trial site, Ageo, Saitama
  - EA Pharma trial site, Iruma, Saitama
  - EA Pharma trial site, Shimotsuga, Tochigi
  - EA Pharma trial site, Bunkyo, Tokyo
  - EA Pharma trial site #1, Minato, Tokyo
  - EA Pharma trial site #2, Minato, Tokyo
  - EA Pharma trial site, Musashino, Tokyo
  - EA Pharma trial site, Shinjuku, Tokyo
  - EA Pharma trial site, tabashi City, Tokyo
  - EA Pharma trial site #1, Fukuoka
  - EA Pharma trial site #2, Fukuoka
  - EA Pharma trial site, Fukushima
  - EA Pharma trial site #1, Hiroshima
  - EA Pharma trial site #2, Hiroshima
  - EA Pharma trial site, Kagoshima
  - EA Pharma trial site, Kumamoto
  - EA Pharma trial site, Kyoto
  - EA Pharma trial site, Niigata
  - EA Pharma trial site, Okayama
  - EA Pharma trial site, Osaka
  - EA Pharma trial site, Saga
  - EA Pharma trial site, Yamagata

IPD SHARING:
Plan to Share IPD: No